CLINICAL TRIAL: NCT01482312
Title: Effect of Contact Lenses on Tear Osmolarity in a Controlled Low Humidity Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-373-C-900
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Myopia; Dry Eye
MeSH Terms: conditions — Myopia; Dry Eye Syndromes | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lotrafilcon A / Comfilcon A / Glasses (Active Comparator): Lotrafilcon A contact lenses worn first, followed by comfilcon A contact lenses, followed by habitual glasses. Each product worn for 90 minutes in a controlled, low-humidity environment (LHE) chamber. Each period separated by a washout of approximately 7 days.
  Interventions: Device: lotrafilcon A contact lenses; Device: comfilcon A contact lenses; Other: Glasses
- comfilcon A / glasses / lotrafilcon A (Active Comparator): Comfilcon A contact lenses worn first, followed by glasses, followed by lotrafilcon A contact lenses. Each product worn for 90 minutes in a controlled, low-humidity environment (LHE) chamber. Each period separated by a washout of approximately 7 days.
  Interventions: Device: lotrafilcon A contact lenses; Device: comfilcon A contact lenses; Other: Glasses
- glasses / lotrafilcon A / comfilcon A (Active Comparator): Glasses worn first, followed by lotrafilcon A contact lenses, followed by comfilcon A contact lenses. Each product worn for 90 minutes in a controlled, low-humidity environment (LHE) chamber. Each period separated by a washout of approximately 7 days.
  Interventions: Device: lotrafilcon A contact lenses; Device: comfilcon A contact lenses; Other: Glasses

INTERVENTIONS:
Device: lotrafilcon A contact lenses — Commercially marketed, silicone hydrogel, single-vision, soft contact lenses FDA-approved for daily and extended (overnight) wear for up to 30 nights of continuous wear.
  Other Names: Air Optix Night and Day AQUA
Device: comfilcon A contact lenses — Commercially marketed, silicone hydrogel, single-vision, soft contact lenses FDA-approved for daily and extended (overnight) wear for up to 30 nights of continuous wear.
  Other Names: Biofinity
Other: Glasses — Glasses per habitual prescription

SUMMARY:
The purpose of this study is to evaluate two different types of contact lenses and their effect on dry eyes when compared to wearing glasses in a controlled, low humidity chamber.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70.
* History of end-of-day or low-humidity dryness with contact lenses.
* Healthy eyes.
* Best-corrected visual acuity of 20/50 or better for each eye.
* Usable pair of eye glasses.
* Willing and able to attend required study visits.
* Sign informed consent.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Ocular or systemic allergies or diseases which might interfere with contact lens wear.
* Clinically significant ocular findings which would contraindicate contact lens wear.
* Unable to abstain from artificial tears or other ophthalmic drops for at least 7 days.
* Participation in another clinical study currently or within 30 days of study entry.
* Spectacle astigmatism of >1.00 diopter.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine participants were randomized into one of three treatment sequences. The study took place at one site, which was located in Canada.
Pre-assignment Details: Participants were instructed to use glasses as a washout from their habitual contact lens brand for at least seven days prior to initiating the first of three LHE (Low-Humidity Environment) chamber visits. This reporting group consists of all enrolled participants.
Period: Period 1, 90 Minutes of Wear
Arm/Group | Lotrafilcon A / Comfilcon A / Glasses | Comfilcon A / Glasses / Lotrafilcon A | Glasses / Lotrafilcon A / Comfilcon A
Started | 10 | 9 | 10
Completed | 9 | 9 | 10
Not Completed | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Period 2, 90 Minutes of Wear
Arm/Group | Lotrafilcon A / Comfilcon A / Glasses | Comfilcon A / Glasses / Lotrafilcon A | Glasses / Lotrafilcon A / Comfilcon A
Started | 9 | 9 | 9 (One participant discontinued between Period 1 and Period 2)
Completed | 8 | 9 | 9
Not Completed | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Period 3, 90 Minutes of Wear
Arm/Group | Lotrafilcon A / Comfilcon A / Glasses | Comfilcon A / Glasses / Lotrafilcon A | Glasses / Lotrafilcon A / Comfilcon A
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled participants.
Arm/Group | Overall
Number analyzed (Participants) | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Tear Osmolarity
Description: The participant spent 90 minutes in the LHE (low humidity environment) chamber, after which tears were sampled from the lower tear meniscus (thin strip of tear fluid at the lower lid margin) and tear osmolarity was measured using a TearLab osmometer, a device that measures the osmolarity of human tears to aid in the diagnosis of dry eye disease. Tear osmolarity is the measure of solid particles (salt) in a solution (tears), and a higher number can be indicative of dry eye disease, while a lower number is generally indicative of the normal tear osmolarity.
Time Frame: 90 minutes
Population: As treated.
Measure: Mean (Standard Deviation); unit: mOsms/L
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon A Contact Lenses | Comfilcon A Contact Lenses | Glasses
Number analyzed (Participants) | 27 | 26 | 27
Number analyzed (Eyes) | 54 | 52 | 54
mOsms/L | 310 (11) | 313 (9) | 306 (11)

2. Primary Outcome: Ocular Comfort
Description: Ocular comfort was assessed by the participant after 90 minutes in the LHE and quantified as a linear measure (cm) on a modified Visual Analog Scale (VAS) of 0-20 cm, with a higher number indicating greater perceived comfort.
Time Frame: 90 minutes
Population: As treated.
Measure: Median (Standard Deviation); unit: cm
Units Other Than Participants: Eyes
Arm/Group | Lotrafilcon A Contact Lenses | Comfilcon A Contact Lenses | Glasses
Number analyzed (Participants) | 27 | 27 | 27
Number analyzed (Eyes) | 54 | 54 | 54
cm | 9.4 (3.98) | 8.2 (3.30) | 9.7 (3.53)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for (duration)
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon A Contact Lenses | Comfilcon A Contact Lenses | Glasses
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.